CLINICAL TRIAL: NCT05059119
Title: Rectovaginal Fistula in Post-Radiotherapy Advanced Cervical Cancer Patients
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 109104-C
Record Dates: First submitted 2021-09-02; First posted 2021-09-28 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced Cervical Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the associated risk factors of rectovaginal fistula

DETAILED DESCRIPTION:
To investigate the associated risk factors of rectovaginal fistula in cervical caner patients after radiotherapy

ELIGIBILITY:
Inclusion Criteria:

Rectovaginal fistula Cervical cancer

Exclusion Criteria:

Nil

Ages: 54 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To present cases who developed rectovaginal fistulas after radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Rate of associated comorbidity or intervention | 12 months
  Rate of associated comorbidity or intervention in patients with rectovaginalfistula

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan